CLINICAL TRIAL: NCT03591510
Title: A Phase II, Open-label, Single Arm Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Twice Daily Midostaurin (PKC412) Combined With Standard Chemotherapy and as a Single Agent Post-consolidation Therapy in Children With Untreated FLT3-mutated AML
Brief Title: A Global Study of Midostaurin in Combination With Chemotherapy to Evaluate Safety, Efficacy and Pharmacokinetics in Newly Diagnosed Pediatric Patients With FLT3 Mutated AML
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPKC412A2218; 2017-004830-28 (EudraCT Number)
Expanded Access: NCT05219266 (No longer available)
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: FLT3-mutated Acute Myeloid Leukemia
Keywords: PKC412; Acute Myeloid Leukemia; AML; FLT3-mutated; pediatric population; midostaurin; midostaurin combined with standard chemotherapy; single agent post-consolidation therapy; untreated FLT3-mutated AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin; fludarabine; Cytarabine; Daunorubicin; Idarubicin; Mitoxantrone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy followed by Midostaurin (Experimental): In Part 1, midostaurin with standard induction (Block 1 induction according to local practice, Block 2 induction containing fludarabine, cytarabine, daunorubicin/idarubicin) and consolidation (Block 3: cytarabine + mitoxantrone, Block 4: cytarabine + etoposide, Block 5: cytarabine) followed by single agent midostaurin post-consolidation therapy.
  In Part 2, midostaurin with standard induction (Block 1 induction according to local practice, Block 2 induction containing cytarabine + mitoxantrone) and consolidation (Block 3: cytarabine + etoposide, Block 4: cytarabine + mitoxantrone, Block 5: cytarabine) followed by single agent midostaurin post-consolidation therapy.
  Interventions: Drug: Midostaurin; Drug: Fludarabine; Drug: Cytarabine; Drug: Daunorubicin or idarubicin; Drug: Mitoxantrone; Drug: Etoposide

INTERVENTIONS:
Drug: Midostaurin — midostaurin 30mg/m2 bid
  Other Names: PKC412
Drug: Fludarabine — 30mg/m2/day on D1-D5 of Block 2 FLADx
  Other Names: Part 1 Block 2 induction FLADx
Drug: Cytarabine — Part 1:
  2000mg/m2/day D1 to D5 of Block 2 FLADx 1000mg/m2 every 12 hours D1 to D3 Block 3 HAM 3000mg/m2 every 12 hours D1 to D3 Block 4 HA3E 3000mg/m2 every 12 hours D1 to D3 Block 5 HIDAC
  Part 2:
  1000mg/m2 every 12 hours D1 to D3 Block 2 HAM 3000mg/m2 every 12 hours D1 to D3 Block 3 HA3E 1000mg/m2 every 12 hours D1 to D3 Block 4 HAM 3000mg/m2 every 12 hours D1 to D3 Block 5 HIDAC
  Other Names: Part 1:; Block 2 induction FLADx; Block 3 consolidation HAM; Block 4 consolidation HA3E; Block 5 consolidation HIDAC; Part 2:; Block 2 induction HAM; Block 3 consolidation HA3E; Block 4 consolidation HAM
Drug: Daunorubicin or idarubicin — daunorubicin 60 mg/m2/day OR idarubicin 12mg/m2/day On D2, D4, D6 of Block 2 FLADx
  Other Names: Part 1 Block 2 induction FLADx
Drug: Mitoxantrone — 10mg/m2/day D3 and D4
  Other Names: Part 1:; Block 3 consolidation HAM; Part 2:; Block 2 induction HAM; Block 4 consolidation HAM
Drug: Etoposide — 100mg/m2/day D1 to D5
  Other Names: Part 1:; Block 4 consolidation HA3E; Part 2:; Block 3 consolidation HA3E

SUMMARY:
This study will evaluate the safety, efficacy and pharmacokinetics of midostaurin in combination with standard chemotherapy in pediatrics patients with newly diagnosed FLT3-mutated Acute Myeloid Leukemia. The study has two parts: Part 1 to define the Recommended Phase 2 Dose, and Part 2 to evaluate safety and tolerability and efficacy of midostaurin. Both parts will consist of 2 induction blocks, 3 consolidation blocks, 12 cycles of post-consolidation consisting of continuous therapy with midostaurin, and a follow-up phase.

DETAILED DESCRIPTION:
This trial is an open label, multi center single arm study to evaluate twice daily oral midostaurin with standard induction, consolidation chemotherapy with sequential midostaurin therapy for 5 treatment blocks (2 induction blocks, 3 consolidation blocks, followed by single agent midostaurin post consolidation therapy for 12 cycles).

The total maximum planned duration on treatment is 17 cycles (5 blocks and 12 cycles). A block is defined as the time from start of study treatment to the time of hematopoietic recovery, at the latest at Day (D) 42, or determination of persistent disease, whichever occur first.

In both Part 1 and Part 2, patients will receive the first course of induction chemotherapy according to local standard and duration is from 8 to 12 days. Upon FLT3 mutation confirmation, patients will receive midostaurin for 14 days. After determination of remission and hematopoietic recovery, patients will receive Block 2.

In Part 1:

* Block 2 FLADx treatment duration is D1 to D6, and midostaurin from D8 to D21. Patients who achieve documented CR (and hematopoietic recovery at the latest at D42 from the first day of Block 2) will receive Block 3.
* Block 3 consolidation HAM treatment duration is D1 to D4, followed by midostaurin D8 to D21. Patients who achieve hematopoietic recovery at the latest at D42 from the first day of Block 3 will receive Block 4. Patients who relapse will discontinue further study treatment.
* Block 4 HA3E treatment duration is D1 to D5 followed by midostaurin D8 to D21. Patients who achieve hematopoietic recovery at the latest at D42 from the first day of Block 4 will receive Block 5.
* Block 5 HiDAC treatment duration is D1 to D3 followed by midostaurin D8 to D21. Patients who relapse will discontinue further study treatment.

Patients in continuous remission with hematopoietic recovery will receive continuous post consolidation therapy of midostaurin, during 12 cycles (28 days per cycle).

In Part 1 of the study, patients in cohorts of 3 will receive sequential midostaurin administered at 30mg/m2bid. If the 30mg/m2 bid is well tolerated as measured by the Dose Limited Toxicity (DLT) rate during Bock 1, additional patients in cohort of 3 will be treated with sequential midostaurin at 60mg/m2 bid. When the recommended phase 2 dose (RP2D) is confirmed, subsequent patients will be treated in Part 2 of the study at the RP2D.

In Part 2:

* Block 2 HAM treatment duration is D1 to D4 and midostaurin from D8 to D21. Patients who achieve documented CR (and hematopoietic recovery at the latest at D42 from the first day of Block 2) will receive Block 3.
* Block 3 consolidation HA3E treatment duration is D1 to D5, followed by midostaurin D8 to D21. Patients who achieve hematopoietic recovery at the latest at D42 from the first day of Block 3 will receive Block 4. Patients who relapse will discontinue further study treatment.
* Block 4 HAM treatment duration is D1 to D4 followed by midostaurin D8 to D21. Patients who achieve hematopoietic recovery at the latest at D42 from the first day of Block 4 will receive Block 5.
* Block 5 HiDAC treatment duration is D1 to D3 followed by midostaurin D8 to D21. Patients who relapse will discontinue further study treatment.

Patients in continuous remission with hematopoietic recovery will receive continuous post consolidation therapy of midostaurin, during 12 cycles (28 days per cycle). Patients who relapse will discontinue further study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented Diagnosis of previously untreated de novo AML according to WHO 2016 criteria
* Presence of a FLT3 mutation status as measured/confirmed by a designated lab with results available prior first dose of Midostaurin
* Patients with Lansky or Karnofsky performance status equal or superior to 60
* Patient with the following laboratory value : AST and ALT ≤ 3times ULN
* Serum Total bilirubin ≤ 1.5times ULN
* Estimated creatinine clearance ≥30ml/min

Exclusion Criteria:

* Any concurrent malignancy, AML with Philadelphia Chromosome, AML-DS, JMML
* Symptomatic leukemic CNS involvement
* Isolated extramedullary leukemia, secondary AML and MDS
* Acute Promyelocytic Leukemia with the PML RARA rearrangement
* Patient who have received prior treatment with a FLT3 inhibitor. However, up to 1 week of FLT3 inhibitor (except midostaurin) exposure prior to study enrollment is permissible.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2029-09-02 (Estimated)

PRIMARY OUTCOMES:
Part 1 of the study: Occurence of dose limiting toxicities (DLT) | From the start of midostaurin treatment in Block 1 to the end of Block 2, from Day 1 to Day 84
  Dose-limiting toxicity (DLT) is defined as any death due to toxicity related to study treatment (chemotherapy + midostaurin) and/or any CTCAE grade 4 non-hematological adverse event or abnormal laboratory value grade 4 related to study treatment unless the event improves sufficiently by day 42 and therefore does not further delay the next cycle of study treatment.
Part 2 of the study: To evaluate Safety of midostaurin (30mg/m2 bid or 1 mg/kg bid for participants <10 kg body weight) in sequential combination with chemotherapy followed by 12 cycles of midostaurin post-consolidation therapy. | From the start of treatment up to 5 years follow-up of last patient
  Safety profile includes type, frequency and severity of adverse events during the induction, consolidation and post consolidation phase. AEs are also collected during post treatment follow-up phase
Part 2 of the study: To evaluate Tolerability of midostaurin (30mg/m2 bid or 1 mg/kg bid for participants <10 kg body weight) in sequential combination with chemotherapy followed by 12 cycles of midostaurin post-consolidation therapy. | From the start of treatment up to 5 years follow-up of last patient
  Number of dose interruptions/reductions and discontinuations due to study drug

SECONDARY OUTCOMES:
Part 2 of the study: Percentage of participants with response (CR, CR/modified CRi and CR/CRi) | From the start of treatment in Block 1 to the end of Block 2, from Day 1 up to Day 84
  Percentage of participants with a response of CR, CRi or modified CRi at the end of Block 2
Part 2 of the study: Time to response (TTR) and response duration | From the start of treatment up to 5 years follow-up of last patient
  TTR is defined as the time between start of treatment to the date of first onset of response (CR, CRi or modified CRi).
  Response duration is defined as the time from CR, CRi or modified CRi to relapse or death due to any cause.
Part 2 of the study: Event Free Survival (EFS) | From the start of treatment to time when all patients have completed at least 18 months of follow up (~ 48 months)
  EFS is defined as the time from Day 1 of chemotherapy until an EFS event is observed.
  An EFS event is defined as a failure to obtain CR/Modified CRi within induction, relapse after CR/modified CRi, or death due to any cause, whichever occurs first. EFS will be measured after all participants completed at least 18 months of follow-up.
Part 2 of the study: Overall Survival (OS) | At each visit, every 3 months after last follow-up visit and up to 5 years after last patient first treatment
  OS is defined as the time from Day 1 of chemotherapy to the date of death due to any cause.
Part 2 of the study: Disease free survival (DFS) | From the start of treatment up to 5 years follow-up of last patient
  DFS is defined as the time from CR/modified CRi in induction to relapse or death due to any cause
Part 2 of the study: Percentage of participants with MRD negative status during each study phase | MRD is evaluated at Day 14 after end of chemotherapy induction Block 1, at Day 21 of Blocks 2, 3, 4 and 5, and Cycle 7 during post-consolidation phase (each block could last up to 42 days)
  Percentage of patient with MRD negative status by multiparameter flow cytometry
Part 2 of the study: Palatability of oral solution of midostaurin | Day 14 after end of chemotherapy induction Block 1, Day 21 of Blocks 2, 3, 4 and 5 (each block can last up to 42 days), post-consolidation Cycle 1, Cycle 3, Cycle 5, Cycle 7, Cycle 9, Cycle 11
  Palatability is assessed through questionnaires- Palatability PRO and obsPRO
Part 2 of the study: Percentage of blasts in bone marrow and peripheral blood | Parameters are assessed 14 days after end of chemotherapy induction Block 1 and Day 14 induction Block 2
  Bone marrow and peripheral blood parameters and extramedullar involvement at the end of induction Block 1 and Block 2
Part 1 and Part 2 of the study: Plasma concentrations of midostaurin and its metabolites | Days 1, 7 & 14 after end of local chemotherapy-induction in Block 1, Days 14 & 21 of Block 2, Day 21 of Blocks 3, 4 & 5 (each block can last up to 42 days), in-post consolidation Day 1 of Cycle (C)2, C3, C5, C7, C9 and C12 (each cycle = 28 days)
  Plasma concentration of midostaurin and its 2 metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Novartis Investigative Site, Prague, Czechia
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
- Italy (4):
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Osaka, Japan
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, Krakow, Poland
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Ljubljana, Slovenia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.